CLINICAL TRIAL: NCT02473068
Title: Non Invasive Ventilation Comfort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CIA-170
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: CPAP

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Group 1 (Active Comparator): In random order, CPAP via a standard humidifier with chamber output temperature of 31°C, or CPAP with a prototype humidifier with chamber output temperature of 31°C.
  Interventions: Device: CPAP
- Group 2 (Experimental): In random order, CPAP via a standard humidifier with chamber output temperature of 31°C, or CPAP with a prototype humidifier with chamber output temperature of 27°C.
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP

SUMMARY:
Patients who are suffering from a variety of respiratory conditions benefit from continuous positive airway pressure (CPAP) which is a form of Non-Invasive Ventilation (NIV). Some patients find the temperature of the breathing gas difficult to tolerate. The aim of this study is to compare comfort of healthy volunteer participants while being given CPAP at different temperatures.

DETAILED DESCRIPTION:
Patients who are suffering from a variety of respiratory conditions benefit from continuous positive airway pressure (CPAP) which is a form of Non-Invasive Ventilation (NIV). Some patients find the temperature of the breathing gas difficult to tolerate. The aim of this study is to compare comfort of healthy volunteer participants while being given CPAP at different temperatures. Healthy volunteers will be given two different levels humidity and temperature and asked about preference.

ELIGIBILITY:
Inclusion Criteria:

* Any employee of FPH willing to take part in the study following review of the Participant Information Sheet and who has provided affirmative answers to the questions / statements included on the Consent Form

Exclusion Criteria:

* Any employee of FPH not willing to take part in the study following review of the Participant Information Sheet.
* Any employee of FPH who has not provided affirmative answers to the questions / statements included on the Consent Form

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Participant Comfort Questionnaire | 30 Minutes
  Participant answers questions to indicate comfort

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Bold, PhD, Principal Investigator — Fisher & Paykel Healthcare
Locations (1):
- Fisher and Paykel Healthcare, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No